CLINICAL TRIAL: NCT07296510
Title: Is it Feasible to Use Data Obtained Through a Three-Dimensional Reconstructed Image to Assist in Prostate Targeted Biopsy?
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ting Huang, Principal Investigator, Zhejiang University
Other Study IDs: 2021120
Record Dates: First submitted 2025-11-23; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate Biopsy

INTERVENTIONS:
Procedure: Prostate biopsy — All participants underwent both targeted and systematic biopsies, along with three-dimensional reconstructed image-assisted prostate targeted biopsy,and software-assisted fusion targeted biopsy

SUMMARY:
Objectives:There are numerous auxiliary methods to improve the accuracy of pathology results regarding prostate biopsy. However, there is no consensus on how to achieve precise targeted biopsy. This paper explores whether using data obtained through the three-dimensional reconstructed image to locate biopsy points can assist in prostate targeted biopsy.

Methods: This study is prospective. Between January 1, 2022, and June 30, 2025, our center conducted prostate biopsies on a total of 436 patients who met the criteria for prostate biopsy and exhibited suspicious lesions (PI-RADS 3-5), totaling 471 lesions. Prior to the biopsies, 3D Slicer software was utilized to perform three-dimensional reconstructions of the pelvic organs. Three-dimensional imaging was employed to measure the biopsy path data, guiding targeted biopsies. This study combined software-assisted targeted biopsies with systematic biopsies and conducted an analysis to assess the feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

Patients meet the criteria for prostate biopsy and exhibited suspicious lesions (PI-RADS 3-5)

Exclusion Criteria:

Patients with advanced prostate cancer and those with severe coagulopathy or other conditions unsuitable for prostate biopsy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participants who presented MRI-visible lesions
Sampling Method: Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
detection rates of clinically significant prostate cancer | 2022.01~2025.06

CONTACTS AND LOCATIONS:
Locations (1):
- Jinhua Hospital, Zhejiang University School of Medicine, Jinhua, Zhejiang, China